CLINICAL TRIAL: NCT03758417
Title: A Phase 2, Open-Label Study of LCAR-B38M CAR-T Cells, a Chimeric Antigen Receptor T-cell (CAR-T) Therapy Directed Against BCMA in Chinese Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of LCAR-B38M CAR-T Cells, a Chimeric Antigen Receptor T-cell (CAR-T) Therapy Directed Against B-cell Maturation Antigen (BCMA) in Chinese Participants With Relapsed or Refractory Multiple Myeloma
Acronym: CARTIFAN-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to a strategic realignment of the sponsor's business plan, not related to safety, efficacy, or data integrity concerns.
Sponsor: Nanjing Legend Biotech Co. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108494; 68284528MMY2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LCAR-B38M Chimeric Antigen Receptor T Cell (Experimental): Participants will receive LCAR-B38M CAR-T cells as a single infusion which consists of autologous T lymphocytes transduced with LCAR-B38M, a lentiviral vector to express a chimeric antigen receptor targeting the human B cell maturation antigen (anti-BCMA CAR).
  In addition, participants will enroll in additional cohort to further characterize the safety profile and accumulate efficacy data of LCAR-B38M CAR-T cells.
  Interventions: Biological: LCAR-B38M CAR-T Cell

INTERVENTIONS:
Biological: LCAR-B38M CAR-T Cell — Participants will receive LCAR-B38M CAR-T cells as a single infusion which consists of autologous T lymphocytes transduced with LCAR-B38M, a lentiviral vector to express a chimeric antigen receptor targeting the human B cell maturation antigen (anti-BCMA CAR).
  Other Names: Ciltacabtagene autoleucel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of LCAR-B38M chimeric antigen receptor T (CAR-T) cells.

ELIGIBILITY:
Inclusion Criteria:

* Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Measurable disease at Screening
* Received at least 3 prior lines of treatment for multiple myeloma

  a) Undergone at least 1 complete cycle of treatment for each line, unless progressive disease (PD) was documented by IMWG criteria as the best response to the regimen
* Received a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD)
* Participant must have documented evidence of progressive disease based on investigator's determination of response consistent with IMWG criteria on or within 12 months of their last regimen. Non-responsive disease is defined as either failure to achieve minimal response or development of progressive disease (PD) while on therapy. Also, participants with documented evidence of PD disease (as above) within the previous 6 months and who are refractory or non-responsive to their most recent line of treatment afterwards are eligible
* Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 or 1

Exclusion Criteria:

* Prior treatment with chimeric antigen receptor T (cells) CAR-T therapy directed at any target
* Any therapy that is targeted to B-cell maturation antigen (BCMA)
* The following cardiac conditions: a) New York Heart Association (NYHA) stage III or IV congestive heart failure b) Myocardial infarction or coronary artery bypass graft (CABG) 6 months prior to enrollment c) History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration d) History of severe non-ischemic cardiomyopathy e) Impaired cardiac function (left ventricular ejection fraction [LVEF] less than [<]45%) as assessed by echocardiogram or multiple-gated acquisition (MUGA) scan (performed less than or equal to (<=) 8 weeks of apheresis)
* Have received a cumulative dose of corticosteroids equivalent to greater than or equal to(>=)70 milligram (mg) of prednisone within 7 days prior to apheresis
* Diagnosed or treated for invasive malignancy other than multiple myeloma, except:

  1. Malignancy treated with curative intent and with no known active disease present for greater than or equal to (>=) 2 years before enrollment; or
  2. Adequately treated non-melanoma skin cancer without evidence of disease
* Prior antitumor therapy with insufficient washout period
* Toxicity from previous anticancer therapy must resolve to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy
* Received either of the following:

  1. An allogeneic stem cell transplant for multiple myeloma
  2. An autologous stem cell transplant less than or equal to (<=) 12 weeks before apheresis
* Known active, or prior history of, central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Minimum 2 years after LCAR-B38M chimeric antigen receptor T (CAR-T) infusion (Day 1)
  The ORR is defined as the percentage of participants who achieve at least a partial response (PR) or better according to international myeloma working group (IMWG) criteria.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Chimeric Antigen Receptor T (CAR-T) Positive Cell Concentration | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Venous blood samples will be collected for measurement of CAR-T positive cellular concentration.
Transgene Levels of LCAR-B38M CAR-T Cells | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Transgene Levels of LCAR-B38M CAR-T Cells using sensitive assay methods will be assessed.
Systemic Cytokine Concentrations | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Serum cytokine concentrations such as Interleukin [IL]-6, IL-15, IL-10 will be measured for biomarker assessment.
Number of Participants With Anti- LCAR-B38M CAR-T Cell Antibodies | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Number of participants with anti- LCAR-B38M CAR-T cell antibodies will be evaluated.
Percentage of Participants with Very Good Partial Response (VGPR) or Better Rate | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  The VGPR or better rate, defined as the percentage of participants achieving VGPR and complete response (CR) (including stringent complete response [sCR]) according to IMWG criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or greater than or equal to (>=) 90 percent (%) reduction in serum Mprotein plus urine M-protein less than (<) 100 milligram (mg)/24 hours, CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells (PCs) in bone marrow. sCR: CR plus normal free light chain (FLC) ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence for 2 to 4 color flow cytometry.
Percentage of Participants with Complete Response (CR) | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Complete response is based on serum M-Protein and bone marrow assessments as per IMWG criteria.
Percentage of Participants with Negative Minimal Residual Disease (MRD) | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Minimal residual disease negative rate is defined as the percentage of participants who achieve MRD negative status by the respective time point. MRD will be assessed by bone marrow 8-colored flow cytometry.
Percentage of Participants who Achieve Clinical Benefit | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Clinical Benefit Rate is defined as the percentage of participants who achieve ORR (sCR + CR + VGPR + PR) and minimal response (MR) as per IMWG criteria.
Duration of Response (DOR) | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Duration of response (DOR) will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria or death due to any cause, whichever occurs first.
Time to Response (TTR) | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Time to response (TTR) is defined as the time between date of the initial infusion of LCAR-B38M CAR-T cells and the first efficacy evaluation that the participant has met all criteria for PR or better.
Progression-Free Survival (PFS) | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  PFS defined as time from date of initial infusion of LCAR-B38M CAR-T cells to date of first documented disease progression, defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Overall survival (OS) | Mnimum 2 years after LCAR-B38M CART infusion (Day 1)
  Overall survival (OS) is measured from the date of infusion of the LCAR-B38M CAR-T cells to the date of the participant's death.
Levels of CAR-T cell Activation Markers | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Levels of CAR-T cell Activation Markers like CD4+, CD8+, and CD25+ will be assessed. An evaluation of cell populations may be performed by flow cytometry.
Levels of LCAR-B38M CAR-T cell Expansion (proliferation) | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Levels of LCAR-B38M CAR-T cell expansion (proliferation) will be reported.
Levels of LCAR-B38M CAR-T Persistence | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Levels of LCAR-B38M CAR-T persistence will be evaluated via monitoring CAR-T positive cell counts and CART transgene levels.
Percentage of Participants with Stringent Complete Response (sCR) | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Stringent Complete Response (sCR) is based on serum M-Protein and bone marrow assessments as per IMWG criteria for complete response(CR) plus normal free light chain (FLC) ratio, and absence of clonal PCs by immunohistochemistry(IHC), or 2 to 4 color flow cytometry.
Circulating Soluble B-Cell Maturation Antigen (sBCMA) Levels | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Blood samples will be collected for measurement of sBCMA level.
Percent Reduction in BCMA Expression Cells | Minimum 2 years after LCAR-B38M CART infusion (Day 1)
  Percent reduction in BCMA Expression Cells will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research&Development,LLC Clinical Trail, Study Director — Janssen Research & Development, LLC
Locations (11):
- China (11):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union hospital, Fuzhou, Fujian
  - Sun Yat -Sen University Cancer Center, Guandong, Guangzhou
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Fourth People Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Medical School of Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Mi JQ, Zhao W, Jing H, Fu W, Hu J, Chen L, Zhang Y, Yao D, Chen D, Schecter JM, Yang F, Tian X, Sun H, Zhuang SH, Ren J, Fan X, Jin J, Niu T, Chen SJ. Phase II, Open-Label Study of Ciltacabtagene Autoleucel, an Anti-B-Cell Maturation Antigen Chimeric Antigen Receptor-T-Cell Therapy, in Chinese Patients With Relapsed/Refractory Multiple Myeloma (CARTIFAN-1). J Clin Oncol. 2023 Feb 20;41(6):1275-1284. doi: 10.1200/JCO.22.00690. Epub 2022 Oct 21. PMID 36269898